CLINICAL TRIAL: NCT06027047
Title: Breakthrough Anxiety and Sleep Evaluation Using Linked Devices and Smartphone Application Onar (BASEL)
Acronym: BASEL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Raivotech (Industry)
Responsible Party: Sponsor
Other Study IDs: ROA101
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Sleep Deprivation; Sleep Hygiene; Sleepiness; Sleep Driving; Depression, Anxiety; Anxiety Disorders; Depressive Symptoms
Keywords: smartphone; wearables; app; sleep; anxiety; depression
MeSH Terms: conditions — Sleep Deprivation; Sleep Hygiene; Sleepiness; Depression; Anxiety Disorders; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sleep is not simply the absence of wakefulness. Sleep is an active procedure, normally happening every night, and is absolutely vital. Good sleep is essential for our well-being. Survival without food can be further than without sleep. Work time and commuting time seem to affect total sleep time and night bedtime. Social and work obligation can, therefore, suppress sleep time. Sleep deprived individuals may be facing anxiety and depression symptoms.

The aim of this study is to investigate the presence of anxiety and depression symptoms among adults with the use of the smartphone application Onar. Onar app will be used to gather information from wearable devices of the users including total sleep time, sleep efficiency, wake after sleep onset time. An established questionnaire (Hospital Anxiety Depression Scale/ HADS) will be used to quantify and detect the presence of anxiety and depression in the study population.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance of terms of use of the application must be done prior to participation in the study.
* Male and female adults aged ≥18 years old and ≤60 years old.
* Subjects using the application on a daily basis for at least 1 week prior to participation.

Exclusion Criteria:

* History of alcohol or other substance abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects using the application on a daily basis for at least 1 week prior to participation will be eligible for participation. After the first full week of data will be over, the application will show a message asking for participation in the study and acceptance of terms.
  Participants will continue using their smartwatch as usual and data will be collected from a period of 2 week for each subject. At the end of the 2-week period a new message will be asking the participant to complete the Hospital Anxiety and Depression Questionnaire (HADS) and the Epworth Sleepiness Scale (ESS) and the total score will be stored.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
To determine the existence of depression and anxiety symptoms in the study population. | 2 weeks
  Comparison of HADS score with population standardized mean value.

SECONDARY OUTCOMES:
Correlation of depression and anxiety symptoms with Total sleep time (TST). | 2 weeks
  Total sleep time (TST).
Correlation of depression and anxiety symptoms with Wake after sleep onset time (WASO). | 2 weeks
  Wake after sleep onset time (WASO).
Correlation of depression and anxiety symptoms with Sleep Onset Latency (SOL). | 2 weeks
  Sleep Onset Latency (SOL).
Correlation of depression and anxiety symptoms with Epworth Sleepiness Scale (ESS). | 2 weeks
  Epworth Sleepiness Scale (ESS).

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakos Karkoulias, Prof., Principal Investigator — University Hospital of Patras, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sforza E, de Saint Hilaire Z, Pelissolo A, Rochat T, Ibanez V. Personality, anxiety and mood traits in patients with sleep-related breathing disorders: effect of reduced daytime alertness. Sleep Med. 2002 Mar;3(2):139-45. doi: 10.1016/s1389-9457(01)00128-9. PMID 14592233
- [Background] Bixler EO, Vgontzas AN, Lin HM, Calhoun SL, Vela-Bueno A, Kales A. Excessive daytime sleepiness in a general population sample: the role of sleep apnea, age, obesity, diabetes, and depression. J Clin Endocrinol Metab. 2005 Aug;90(8):4510-5. doi: 10.1210/jc.2005-0035. Epub 2005 Jun 7. PMID 15941867
- [Background] Horenstein A, Morrison AS, Goldin P, Ten Brink M, Gross JJ, Heimberg RG. Sleep quality and treatment of social anxiety disorder. Anxiety Stress Coping. 2019 Jul;32(4):387-398. doi: 10.1080/10615806.2019.1617854. Epub 2019 May 13. PMID 31082285
- [Background] Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003 Aug 1;1:29. doi: 10.1186/1477-7525-1-29. PMID 12914662